CLINICAL TRIAL: NCT02469376
Title: Biodistribution, Imaging Properties, and Radiation Dosimetry of [18F]-GP1 Positron Emission Tomography (PET) Tracer in Vascular Disease Imaging
Brief Title: Evaluation of a New Imagingtechnologie for Thrombosis
Acronym: PET-GP1_1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: University of Zurich (Other)
Collaborators: Life Molecular Imaging SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PET - GP1_1
Record Dates: First submitted 2015-06-08; First posted 2015-06-11 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Abdominal Aortic Aneurysm; Deep Vein Thrombosis
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnosis with GP1 (Experimental): Injection and scanning of [18F]-GP1
  Interventions: Drug: [18F]-GP1

INTERVENTIONS:
Drug: [18F]-GP1 — Radiopharmaceutical Product (Tracer) to visualize with Positron Emission Tomography a thrombus in humans.
  Other Names: GP1

SUMMARY:
Arterial and venous thrombi play an important role in various vascular diseases such as myocardial infarction, stroke, transient ischemic attacks (TIA) and pulmonary embolism. These thromboembolic disorders are the leading causes of morbidity and mortality worldwide. A non-invasive method for the quantitative and effective detection of thrombi in the whole body has not yet been established. In spite of the available techniques, 30% to 40% of ischemic strokes "cryptogenic" (undetermined cause, the source of thromboembolism is never identified). Possible causes of cryptogenic stroke atherosclerosis include in the aortic arch or intracranial arteries. A plaque in the arch or other large vessels could be an important source of cryptogenic strokes, however, are those difficult to detect by routine methods. The approach of thrombus targeted molecular imaging could identify potentially troublesome plaques early on before they become a dangerous rupture. The hypothesis is that the radiotracer 18F-arterial GP1 and venous thrombi using positron emission tomography (PET) can be made visible. The primary goal is the potential applicability of the substance as a PET tracer for diagnosing thrombi.

DETAILED DESCRIPTION:
This is a first in man study with which we are testing the feasibility of the use of this radiopharmaceutical product to visualize a thrombus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AAA (diameter >3.5cm in duplex sonography) or acute DVT.
* Male and female patients 18 years and older,
* Signed Informed Consent after being informed

Exclusion Criteria:

* contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product,
* women who are pregnant or breast feeding,
* women with the intention to become pregnant during the course of the study,
* other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease),
* renal clearance < 30 mL/min
* known or suspected non-compliance, drug or alcohol abuse,
* inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the subject,
* participation in another study with an investigational drug during the present study and 7 days thereafter.
* enrolment of the investigator, his family members, employees and other dependent persons
* last systemic treatment with GP IIb/IIIa antagonists should not have been applied within 48 h before performing study exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Assessment of biodistribution of [18F]-GP1 and its properties as a PET imaging agent for detection of abdominal aortic aneurysm (AAA) and deep vein thrombosis (DVT). | 12 Months
  Biodistribution and diagnostic properties of the new Tracer

SECONDARY OUTCOMES:
Calculation of the effective dose to the patient according to the tissue distribution data of [18F]-GP1 (Dosimetry) | 12 Months
  Dosimtery assessment of the new Tracer

CONTACTS AND LOCATIONS:
Overall Officials: Philipp A Kaufmann, Prof, Principal Investigator — University Hospital Zurich, Department of Nuclear Medicine
Locations (1):
- University Hospital Zurich, Division of Nuclear Medicine, Zurich, Canton of Zurich, Switzerland